CLINICAL TRIAL: NCT03225924
Title: Phase Ib - II Study of Entospletinib (ENTO) in Newly Diagnosed Diffuse Large B Cell Lymphoma (DLBCL) Patients With aaIPI>=1 Treated by Rituximab, Cyclophosphamide, Hydroxydaunomycin, Oncovin, and Prednisone (R-CHOP)
Brief Title: Study of Entospletinib (ENTO) in Newly Diagnosed DLBCL Patients With aaIPI>=1 Treated by Chemiotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Stop of drug development
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENTO-R-CHOP
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: DLBCL
MeSH Terms: interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Entospletinib + Rituximab + Cyclophosphamide + Doxorubicine + Vincristine + Prednisone
  Interventions: Drug: Entospletinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Entospletinib — 200mg or 400mg twice a day for 7 days every 21 cycles - total of 8 cycles
  Other Names: ENTO
Drug: Rituximab — cycles of 21 days - 375mg/m²
  Other Names: Mabthera
Drug: Cyclophosphamide — cycles of 21 days - 750 mg/m²
Drug: Doxorubicin — cycles of 21 days - 50mg/m²
Drug: Vincristine — cycles of 21 days - 1.4mg/m²
Drug: Prednisone — cycles of 21 days - 40mg/m²

SUMMARY:
The primary objective of the phase Ib of the study is to determine the recommended phase 2 dose (RP2D) for entospletinib (ENTO) in patients treated with R-CHOP.

The primary objective of the phase II is to determine the complete metabolic response (CMR) rate by the Lugano classification 2014 (Deauville scale 1-3) at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed de novo DLBCL (CD20 positive) (cf section 20.6 - Appendix 4)
2. Age between 60 and 80 years included, on the day of the informed consent document signature
3. Age adjusted International Prognosis Index (aaIPI) score ≥ 1
4. No prior treatment for DLBCL. However prephase treatment with 1mg/kg/day prednisone or equivalent, for a maximum of 14 days, is permitted prior to begin the treatment
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (0 or 1 only for phase 1b)
6. Life expectancy of ≥ 90 days (3 months) before starting Entospletinib
7. Signed informed consent
8. At least one bi-dimensionally measurable lesion defined as at least one node or tumor lesion on CT scan ≥ 1.5 cm
9. fluorodeoxyglucose (FDG) positron emission tomography (PET-CT) performed at baseline with a FDG positive result
10. Adequate hematologic functions defined as follows (unless secondary to bone marrow involvement by lymphoma):

    * Absolute neutrophil count (ANC) > 1.5 X 10^9 G/l and
    * Platelets count ≥ 75 X 10^9/l without platelet transfusion dependency during the last 7 days and
    * Haemoglobin level > 9 g/dl (may receive transfusion)
11. Adequate liver function defined as follows:

    * Total bilirubin <1.5 upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome and
    * Alkaline phosphatase (in absence of bone disease), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 X ULN
12. Adequate renal function as calculated by a creatinine clearance > 40 ml/min by local institutional formula
13. Patients with prior Hepatitis B must be given antiviral prophylaxis and hepatitis B virus (HBV) DNA monitored; Patients with prior Hepatitis C are eligible if, hepatitis C virus (HCV) RNA is undetectable.
14. Left ventricular ejection fraction (LVEF) ≥ 50% of echocardiography or multiple gated acquisition (MUGA) scan
15. Adequate tissue for central retrospective testing for cell of origin (10-15 slides of tumor biopsy must be available at baseline)
16. Heterosexually active females of childbearing potential (as defined in the protocol) must:

    * have a negative serum pregnancy test at baseline and prior to the first study drug administration (C1D-4)
    * have practiced at least 1 reliable method of contraception for at least 2 months prior to the first study drug administration (C1D-4)
    * agree to utilize highly effective methods of contraception (as defined in the protocol) from Cycle 1 Day -4 until 12 months following the last treatment administration
17. Heterosexually active males with partners of childbearing potential must agree to use reliable forms of contraception during treatment and up to 12 months after last treatment administration
18. Male subjects must agree to avoid sperm donation from Cycle 1 Day -4 until 12 months following the last treatment administration

Exclusion Criteria:

1. Central nervous system or meningeal involvement with DLBCL
2. Contraindication to any drug contained in the chemotherapy regimen
3. Prior treatment with Entospletinib or other spleen tyrosine kinase (SYK ) inhibitor
4. Patients with a prior history of other malignancy, exceptions include:

   * a subject who has been disease-free after curative local treatment (surgical resection) for at least 3 years,
   * a subject with a history of a completely resected non-melanoma skin cancer or in situ carcinoma with surgical complete excision.
5. Patients taking current therapy with proton pump inhibitors and current therapy with medicines that are strong Cytochrome P450 3A (CYP3A) or CYP2C9 inducers, or moderate CYP2C9 inducers.
6. Ongoing active pneumonitis
7. Peripheral sensory or motor neuropathy grade > 1.
8. Major surgery within 4 weeks before first dose of study drug (minor procedures including transcutaneous biopsy, central line placement are permitted at any time)
9. Inability to take oral medication or malabsorption syndrome or any other uncontrolled gastrointestinal condition that would impair ability to take entospletinib
10. Significant cardiovascular impairment: congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of first dose of entospletinib or ventricular arrhythmia
11. Active infection as judged by the investigator
12. Known hypersensitivity to ENTO
13. Congenital immunodeficiency or known HIV (human immunodeficiency virus infection) or active viral hepatitis B or C
14. Any other major illness that in the investigator's judgement, will substantially increase the risk associated with the subject's participation in the study
15. Subjects who have undergone a solid organ transplant and stem cell transplant
16. Previous treatment for B cell lymphoma or Richter's transformation
17. Primary Mediastinal B Cell Lymphoma

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Phase I: recommended phase 2 dose | 6 months
  To determine the recommended phase 2 dose for Entospletinib
Phase II: Complete Metabolic Response (CMR) rate at the end of treatment | 168 days
  To determine the CMR rate by the Lugano classification 2014 (Deauville scale 1-3) at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Salles, Principal Investigator — Hospices Civils de Lyon; Emmanuelle Tchernonog, Principal Investigator — University Hospital, Montpellier; Julien Depaus, Principal Investigator — UCL Namur
Locations (27):
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Clinique Universite Catholique de Louvain Saint-Luc, Brussels
  - University Hospital Gent, Ghent
  - Hopital Joliment, Haine-Saint-Paul
  - Az Groeninge, Kortrijk
  - UCL Namur, Yvoir
- France (21):
  - Ch de Bourg En Bresse, Bourg-en-Bresse
  - CHU Côte de Nacre, Caen
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Ch de Versailles - Hopital Andre Mignot, Le Chesnay
  - Clinique Victor Hugo, Le Mans
  - Chu de Limoges - Hopital Dupuytren, Limoges
  - Clinique de La Sauvegarde, Lyon
  - CHU Lyon Sud, Lyon
  - CHU Montpellier, Montpellier
  - Ch Region Mulhouse Et Sud Alsace, Mulhouse
  - Hopital Necker Paris, Paris
  - Chu de Bordeaux, Pessac
  - Ch Annecy Genevois, Pringy
  - Chu de Reims - Hopital Robert Debre, Reims
  - Chu de Rennes - Pontchaillou, Rennes
  - Ch de Roubaix-Hopital Victor Provo, Roubaix
  - Iuct Oncopole de Toulouse, Toulouse
  - Hôpital Bretonneau- Centre H. Kaplan, Tours
  - Ch de Valenciennes, Valenciennes
  - Chru de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No